CLINICAL TRIAL: NCT04490733
Title: Developing Risk Prediction Model of Mild Cognitive Impairment in Patients With Colorectal Cancer From Active Treatment to Survivor and Testing the Effect of Dual Task Walking on Improving Cognitive Function
Brief Title: Developing Risk Prediction Model and Testing the Effect of Dual Task Walking on Improving Cognitive Function in Patients With Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 201912231RINC
Record Dates: First submitted 2020-07-26; First posted 2020-07-29 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; cognitive impairment; chemotherapy; dual-task walking; surgery
MeSH Terms: conditions — Colorectal Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group will receive 3 times interventions during chemotherapy and 12 weekly phone calls or via LINE to assess barriers of dual-task walking.
  Interventions: Behavioral: dual-task walking
- Control group (No Intervention): Participants in control group will receive usual care.

INTERVENTIONS:
Behavioral: dual-task walking — Participants in the experimental group will receive 3 times interventions during chemotherapy and 12 weekly phone calls or via LINE to assess barriers of dual-task walking.
  Arms: Experimental group

SUMMARY:
The aims of this three-year study are to explore cognitive function under different stages of colorectal cancer (CRC) and its related factors; and understand its disturbance and coping process caused by cancer-induced cognitive impairment (CICI) from patient perspective; and further to test effect of dual-task walking on improving cognitive function in CRC patients.

DETAILED DESCRIPTION:
In the first phase, a cross-sectional design will be used to explore both subjective and objective cognitive functions under different cancer treatment trajectories of CRC and their related factors. Additionally, a risk prediction model for mild cognitive impairment will be developed by examining the effects of surgery and chemotherapy on cancer-induced cognitive impairment (CICI) , with the aim of identifying high-risk populations. A qualitative design will be employed to understand the disturbances and coping processes caused by CICI from the patient's perspective. A longitudinal design will be used to examine the effects of surgery and chemotherapy on cognitive function. In the second phase, we will develop a dual-task walking training program and use a randomized controlled trial to test its effect on improving cognitive function (memory, executive function, and attention) in CRC patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed stage I to III colorectal cancer.

Exclusion Criteria:

* Patients with cancer other than colorectal cancer or have cancer recurrence.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-report Questionnaire | In the cross-sectional design, data will be collected at a one-time point; in the longitudinal design and the randomized controlled trial, data will be collected at baseline and 3, 6, and 12 months follow-up.
  The questionnaires include (1) 37 items to assess perceived cognitive functioning and (2) 6 items to assess perceived cognitive impairment.
Neuropsychological test battery | In the cross-sectional design, data will be collected at a one-time point; in the longitudinal design and the randomized controlled trial, data will be collected at baseline and 3, 6, and 12 months follow-up.
  A battery of neuropsychological tests will be used to assess cognitive domains of executive function.
Neuropsychological test battery | In the cross-sectional design, data will be collected at a one-time point; in the longitudinal design and the randomized controlled trial, data will be collected at baseline and 3, 6, and 12 months follow-up.
  A battery of neuropsychological tests will be used to assess cognitive domains of attention.
Neuropsychological test battery | In the cross-sectional design, data will be collected at a one-time point; in the longitudinal design and the randomized controlled trial, data will be collected at baseline and 3, 6, and 12 months follow-up.
  A battery of neuropsychological tests will be used to assess cognitive domains of memory.

SECONDARY OUTCOMES:
Self-report Questionnaire | In the cross-sectional design, data will be collected at a one-time point; in the longitudinal design and the randomized controlled trial, data will be collected at baseline and 3, 6, and 12 months follow-up.
  The questionnaire includes 24 items to assess symptom severity

OTHER OUTCOMES:
Self-report Questionnaire | In the cross-sectional design, data will be collected at a one-time point; in the longitudinal design and the randomized controlled trial, data will be collected at baseline and 3, 6, and 12 months follow-up.
  The questionnaire includes 15 items to assess fatigue level
Self-report Questionnaire | In the cross-sectional design, data will be collected at a one-time point; in the longitudinal design and the randomized controlled trial, data will be collected at baseline and 3, 6, and 12 months follow-up.
  The questionnaire includes 20 items to assess depressive symptom

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ching Shun, PHD, Study Chair — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang HY, Chang YL, Lin BR, Chou YJ, Shun SC. Cognitive Function in Patients at Different Stages of Treatment for Colorectal Cancer: A Comparative Cross-Sectional Study. Semin Oncol Nurs. 2023 Aug;39(4):151446. doi: 10.1016/j.soncn.2023.151446. Epub 2023 May 13. PMID 37183103